CLINICAL TRIAL: NCT00065000
Title: Impact of Non-Commercialism Policy in Seattle Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: DK63899 (completed)
Record Dates: First submitted 2003-07-16; First posted 2003-07-18 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Water

INTERVENTIONS:
Behavioral: Water, Cafeteria and Staff Health Promotion

SUMMARY:
This is a 3-year pilot study funded by National Institute of Health will assess and evaluate obesity-related health outcomes of a real-life policy decision, recently voted on and adopted by the Seattle School Board.

ELIGIBILITY:
Inclusion: All students who attend Cleveland and Rainier Beach high schools are eligible.

Exclusion: Those who are no longer attending those schools.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Dates: Study Completion 2003-08

CONTACTS AND LOCATIONS:
Overall Officials: Donna Johnson, RD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- See also: Center for Public Health Nutrition at University of Washington — http://depts.washington.edu/uwcphn